CLINICAL TRIAL: NCT04919850
Title: Effect of 60-days Saccharomyces Boulardii and Superoxide Dismutase Supplementation on Body Composition, Hunger Sensation, Pro/Antioxidant Ratio, Inflammation and Hormonal Lipo-metabolic Biomarkers in Obese Adults: a Double-blind, Placebo-controlled Trial
Brief Title: Effect of 60-days Saccharomyces Boulardii and Superoxide Dismutase Supplementation in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Principal Investigator, Mariangela Rondanelli, Professor, Azienda di Servizi alla Persona di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1209/151217
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Superoxide Dismutase
MeSH Terms: conditions — Obesity | interventions — Superoxide Dismutase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): A complex of 250 mg of Saccharomyces boulardii and 500 IU SOD to be assumed twice/day for 8 weeks at mealtimes
  Interventions: Dietary Supplement: Saccharomyces boulardii and SOD
- Placebo group (Placebo Comparator): A placebo consisting of capsules containing the same excipients except the active compounds, and the same coating
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces boulardii and SOD — A complex of 250 mg of Saccharomyces boulardii and 500 IU SOD to be assumed twice/day for 8 weeks at mealtimes
  Arms: Intervention group
Combination Product: Placebo — A placebo consisting of capsules containing the same excipients except the active compounds, and the same coating
  Arms: Placebo group

SUMMARY:
In animals it has been demonstrated that Saccharomyces boulardii decrease low-grade inflammation and fat mass; also Superoxide Dismutase (SOD) decrease low-grade inflammation. Therefore, the aim of this double-blind, placebo-controlled clinical trial was to assess the effect of a 60-days S. boulardii and SOD supplementation on circulating markers of inflammation, body composition, hunger sensation, pro/antioxidant ratio, hormonal, lipid profile, glucose, insulin and HOMA-IR, in obese adults (BMI 30-35 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* I class of obesity (BMI: 30-35 Kg/m2)

Exclusion Criteria:

* evidence of heart, kidney or liver disease
* diagnosis of major depressive disorder
* current medications for weight loss, for control of cholesterol and triglycerides
* anti-inflammatory treatments
* pregrancy of lactation
* type 1 diabetes mellitus, intestinal inflammatory bowel disease, celiac disease, chronic pancreatitis
* probiotic/prebiotic treatment in the last 4 weeks
* antibiotic use within the last 3 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Change on concentration of biochemical parameters for hunger sensation and hormonal status | Changes from baseline biochemical parameters for hunger sensation and hormonal status at 8 weeks
  Ghrelin (pg/mL), Adiponectin (pg/ml), Peptide YY (pg/ml)
Change on concentration of biochemical parameters for hunger sensation and hormonal status | Changes from baseline biochemical parameters for hunger sensation and hormonal status at 8 weeks
  Leptin (ng/cL)
Change on concentration of biochemical parameters for hunger sensation and hormonal status | Changes from baseline biochemical parameters for hunger sensation and hormonal status at 8 weeks
  glucagon-like peptide - 1 (pmol/L)
Change on concentration of biochemical parameters for glico-metabolic status | Changes from baseline biochemical parameters for glico-metabolic status at 8 weeks
  Total cholesterol (mg/dL), Low Density Lipoprotein cholesterol (mg/dL), HDL cholesterol (mg/dL), Triglycerides (mg/dL), Apolipoprotein A (mg/dL), Apolipoprotein B (mg/dL), Glycemia (mg/dL), Uric acid (mg/dL)
Change on concentration of biochemical parameters for glico-metabolic status | Changes from baseline biochemical parameters for glico-metabolic status at 8 weeks
  Insulin (mcU/mL)
Change on concentration of biochemical parameters for glico-metabolic status | Changes from baseline biochemical parameters for glico-metabolic status at 8 weeks
  Total Proteins (g/dL), Albumin (g/dL)
Change on concentration of biochemical parameters for glico-metabolic status | Changes from baseline biochemical parameters for glico-metabolic status at 8 weeks
  HOMA index (pt)
Change on state of hunger, fullness, desire to eat, satiety and prospective food consumption | Changes from baseline state of hunger, fullness, desire to eat, satiety and prospective food consumption at 8 weeks
  Eating motivation Visual Analogue Scale (pt): a scale from 0 to 10 points. The scale of hunger (question: "how hungry are you?") ranged from the answer "not at all" to "as hungry as I have ever felt"; the scale of fullness (question: "how full are you?") ranged from the answer "not at all" to "as full as I ever felt"; the scale of satiety (question: "how satiated are you?") ranged from "not at all" to "extremely"; the scale of desire (question: "how strong is your desire to eat?") ranged from "very weak" to "very strong"; the scale of prospective consumption (question: "how much do you think you could (or would want to) eat right now) ranged from "nothing at all" to "a very large amount"

SECONDARY OUTCOMES:
Change on concentration of biochemical parameters for nutritional status | Changes from baseline biochemical parameters for nutritional status at 8 weeks
  Iron (µg/dL)
Change on concentration of biochemical parameters for hormonal status | Changes from baseline biochemical parameters for hormonal status at 8 weeks
  Thyroid Stimulating Hormone (µU/dL)
Change on concentration of biochemical parameters for inflammation and cardiovascular risk | Changes from baseline biochemical parameters for inflammation and cardiovascular risk at 8 weeks
  C-Reactive Protein (mg/dL)
Change on concentration of biochemical parameters for inflammation and cardiovascular risk | Changes from baseline biochemical parameters for inflammation and cardiovascular risk at 8 weeks
  Tumor Necrosis Factor-α (pg/mL), Inter Leukin-1β (pg/mL), Inter Leukin-6 (pg/mL)
Change on concentration of biochemical parameters for inflammation and cardiovascular risk | Changes from baseline biochemical parameters for inflammation and cardiovascular risk at 8 weeks
  Trimethylamine (µM), Trimethylamine-N-oxide (µM)
Change on concentration of biochemical parameters for safety | Changes from baseline biochemical parameters for safety at 8 weeks
  Aspartate amino transferase (U/L), Alanine amino transferase (U/L), Gamma Glutamyl Transferase (U/L)
Change on concentration of biochemical parameters for safety | Changes from baseline biochemical parameters for safety at 8 weeks
  Creatinine (mg/dl)
Change on rate of anthropometric measures | Changes from baseline anthropometric measures at 8 weeks
  Height (cm), waist circumference (cm)
Change on rate of anthropometric measures | Changes from baseline anthropometric measures at 8 weeks
  Weight (Kg)
Change on rate of anthropometric measures | Changes from baseline anthropometric measures at 8 weeks
  Body mass index (kg/m2)
Change on rate of body composition | Changes from baseline body composition at 8 weeks
  Free Fat Mass (kg), Fat Mass (kg)
Change on rate of body composition | Changes from baseline body composition at 8 weeks
  Android fat (%), Gynoid fat (%)
Change on rate of body composition | Changes from baseline body composition at 8 weeks
  Visceral Adipose Tissue (g)
Change on status of mood assessment | Changes from baseline mood assessment at 8 weeks
  Beck questionnaire (pt). The questionnaire is divided into 21 items which have a score from 0 to 3. A total score > 17 indicates borderline depression; > 21 moderate depression; > 31 severe depression; > 40 extreme depression.
Change on status of assessment of food preferences | Changes from baseline assessment of food preferences at 8 weeks
  Food Frequency Questionnaire (pt). Participants must indicate the consumption of 18 common food items, choosing one between "yes" or "no, never". Participants were also asked to estimate their usual rate of consumption, choosing from seven categories of frequency, ranging from ''never'' or ''less than once a week'' to ''seven times per week". The only exception was constituted by the item "coffee consumption", which is reported as "cups/day".

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No